CLINICAL TRIAL: NCT01183819
Title: Cognitive Control and Physical Exercise: A Multi-Modal Intervention
Brief Title: Cognitive Control and Physical Exercise
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Yaakov Stern, Professor of Clinical, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AAAE5848; R01AG034178 (NIH)
Record Dates: First submitted 2010-08-16; First posted 2010-08-18 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Cognitive Function; Day-to-Day Function
Keywords: cognitive function; fMRI; apoE; inflammatory markers; exercise; cognitive intervention; Space Fortress
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Space Fortress and Exercise (Experimental): Participants engage in aerobic exercise 4 times week and Space Fortress sessions 3 times a week for a total of 12 weeks.
  Interventions: Behavioral: Space Fortress; Behavioral: Aerobic Exercise
- Control Games and Exercise (Active Comparator): Participants engage in aerobic exercise 4 times a week and control game sessions 3 times a week for a total of 12 weeks.
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Control Games
- Control Games and Stretching (Active Comparator): Participants engage in stretching/toning exercises 4 times a week and control game sessions 3 times a week for a total of 12 weeks.
  Interventions: Behavioral: Stretching; Behavioral: Control Games

INTERVENTIONS:
Behavioral: Space Fortress — Space Fortress sessions 3 times a week for 12 weeks
  Arms: Space Fortress and Exercise
Behavioral: Aerobic Exercise — Aerobic Exercise 4 times a week for 12 weeks
  Arms: Control Games and Exercise; Space Fortress and Exercise
Behavioral: Stretching — Stretching/Toning exercise 4 times a week for 12 weeks.
  Arms: Control Games and Stretching
Behavioral: Control Games — Control games session 3 times a week for 12 weeks
  Arms: Control Games and Exercise; Control Games and Stretching

SUMMARY:
The purpose of this study is to test the hypothesis that aerobic exercise and a computer-based cognitive intervention leads to improved cognitive function accompanied by increases in gray matter density and changes in functional magnetic resonance imaging (fMRI) patterns of task-related activation.

DETAILED DESCRIPTION:
Epidemiological evidence suggest that a set of lifetime exposures including educational and occupational attainment and leisure activities later in life are associated with more preserved cognitive and day-to-day functioning and reduced risk of dementia. However, the specific set of activities that can maintain or improve function in late life are relatively unexplored. In the current study, we will test the combined efﬁcacy of two such activities: cognitive training and aerobic exercise. These activities have been shown to increase cognitive function and brain plasticity, respectively. The cognitive intervention that we will use is training with the Space Fortress task. This task is aimed at improving cognitive control processes that underlie multiple activities and are particularly affected by aging. We hypothesize that combining these two interventions will produce synergistic effects that will signiﬁcantly improve cognitive and day-to-day function in healthy older adults.

A total of 90 cognitively-healthy older adults will be recruited and randomly assigned to one of three conditions: control video game, control exercise and combined exercise and space fortress training. A range of cognitive and day-to-day functioning will be assessed at baseline and after three months of training. We will also assess compliance with a home-based version of the training program from the end of the 3-month laboratory-based training and the effect of this compliance on measures of cognition and day-to-day functioning. We hypothesize that the interventions can be sustained over a 1-year period and that larger beneﬁts will be observed in participants that adhere to the protocol.

We also propose two complementary approaches to investigating the neural correlates of the beneficial effects of aerobic exercise on cognition: 1) imaging -- we will use a combination of structural, metabolic, and cognitive activation fMRI studies to evaluate the neural substrates of the effect of aerobic exercise on cognition. 2) important correlates -- we will explore the effects of apolipoprotein E (APOE) genotype, inflammatory markers and cognitive reserve on the cognitive effects of aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60-75
2. English-speaking
3. Strongly right-handed
4. BMI > 18.5 and < 32
5. Post-menopausal (women only): no estrogen replacement therapy
6. Sedentary: VO2max < 36 ml/kg/min for men age 60-75; < 29 ml/kg/min for women age 60-75 (determined using Jones Formula Men = (60-(0.55*AGE)) Women = (48-(.37*AGE))

Exclusion Criteria:

1. MRI contraindications (e.g., metallic implants, pacemaker, weight > 350 lbs, waist > 55")
2. Hearing impaired/hearing aids, unable to read newspaper at arm's length with corrective lenses
3. Objective cognitive impairment
4. Ischemic changes, abnormal blood pressure responses, or any significant ectopy during aerobic capacity testing
5. Cardiovascular disease
6. Uncontrolled high blood pressure (systolic blood pressure ≥ 180 mmHg; or diastolic blood pressure ≥ 105 mmHg on two measures)
7. Current or recent (evidence of disease x 5 years) non-skin neoplastic disease or melanoma
8. Active hepatic disease (not a history of hepatitis) or primary renal disease requiring dialysis, primary untreated endocrine diseases, e.g., Cushing's disease or primary hypothalamic failure or insulin dependent diabetes (Type I or II).
9. HIV infection
10. Pregnant or lactating (participation allowed 3 months after ceasing lactation
11. Other medical disorders judge to interfere with study
12. Medications that target CNS (e.g., neuroleptics, anticonvulsants, antidepressants, benzodiazepines) within the last month
13. Women: any selective estrogen receptor modulator or aromatase inhibitor Men: androgen ablation/deprivation hormonal therapies
14. Any history of psychosis or electroconvulsive therapy
15. Psychotic disorder (lifetime)
16. Current or recent (within past 12 months) alcohol or substance abuse or dependence. Recent use (past month) of recreational drugs.
17. Brain disorder such as stroke, tumor, infection, epilepsy, multiple sclerosis, degenerative diseases, head injury, mental retardation
18. Imaged cortical stroke or large subcortical lacunae or infarct or space-occupying lesion (≥ 2 cubic cm). Other findings, e.g., periventricular caps or small white matter hyperintensities, do not result in exclusion
19. Diagnosed learning disability, dyslexia

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in measures of executive control function and episodic memory at 6 months | Baseline and 12 weeks
  tests of global intelligence, executive function, working memory and processing speed

SECONDARY OUTCOMES:
Changes in brain structure, resting cerebral blood flow and network efficiency at 6 months | Baseline and 12 weeks
  structural MRI (for gray matter density), resting CBF (arterial spin labeling) and cognitive activation fMRI studies
Change in aerobic capacity at 6 months | Baseline and 12 weeks
  aerobic capacity as measured by VO2 max
Changes in measures of executive control function and episodic memory at 1 year | Baseline and 52 weeks
  tests of global intelligence, executive function, working memory and processing speed

CONTACTS AND LOCATIONS:
Overall Officials: Yaakov Stern, Ph.D., Principal Investigator — Sergievsky Center Columbia University Medical Center; Richard Sloan, Ph.D., Principal Investigator — Behavioral Medicine Columbia University Medical Center
Locations (1):
- Columbia University Medical Center, New York, New York, United States